CLINICAL TRIAL: NCT03421548
Title: Intraocular Pressure Monitoring With Implantable Intraocular Pressure Sensor for Improved Glaucoma Monitoring in Patients With Boston Keratoprosthesis Type 1
Brief Title: Implantable Intraocular Pressure Sensor for Glaucoma Monitoring in Patients With Boston Keratoprosthesis Type 1
Acronym: BKPro
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The product company withdrawn interest in participation in this study
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Implandata Ophthalmic Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6261
Record Dates: First submitted 2017-08-01; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2016-04

CONDITIONS: Glaucoma; Blindness, Acquired; Keratitis, Herpetic; Ocular Cicatricial Pemphigoid; Corneal Injuries; Corneal Disease; Corneal Opacity
MeSH Terms: conditions — Glaucoma; Blindness; Keratitis, Herpetic; Pemphigoid, Benign Mucous Membrane; Corneal Injuries; Corneal Diseases; Corneal Opacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BKpro I with EyeMate (Experimental): Keratoprosthesis surgery indicated, defined as having a severely opaque and vascularised cornea AND either a verifiable history of two or more prior failed corneal transplant procedures, limbal stem cells deficiency or a medical condition such as alkali burns or autoimmune disease that makes the success of a traditional corneal transplant procedure unlikely. Potential study subjects will be solicited for participation in the clinical trial only after they have consented to the keratoprosthesis operation.
  Interventions: Device: EyeMate
- BKpro I (No Intervention): Keratoprosthesis surgery indicated, defined as having a severely opaque and vascularised cornea AND either a verifiable history of two or more prior failed corneal transplant procedures, limbal stem cells deficiency or a medical condition such as alkali burns or autoimmune disease that makes the success of a traditional corneal transplant procedure unlikely. Potential study subjects will be solicited for participation in the clinical trial only after they have consented to the keratoprosthesis operation.

INTERVENTIONS:
Device: EyeMate — Patients will undergo implantation BKPro with concomitant implantation of the EyeMate pressure sensor. The surgical approach will involve a trephination of the central recipient cornea of adequate size. In subjects with adequate capsular support, the sensor device will be placed in the sulcus space by grasping the sensor's silicone sleeve at approximately the 3 and 9 o'clock positions and sliding it into the sulcus space. In subjects in whom capsular support is inadequate, the Eyemate implant will be sutured to the sclera. This is performed by placing an 8-O Gortex suture or 9-O prolene on CIF-4 needles around the antenna at the 2 and 7 o'clock positions and suturing the device to the sclera using an ab-interno technique.
  Arms: BKpro I with EyeMate

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the EYEMATE system in patients undergoing concomitant implantation of a BKPro type 1 and an EYEMATE sensor over the 24 months period beginning at implantation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of the EYEMATE system in patients undergoing concomitant implantation of a BKPro type 1 and an EYEMATE sensor over the 24 months period beginning at implantation. The EYEMATE system involves an EYEMATE implantable sensor working together with a MESOGRAPH hand-held reading device. The aim of this investigation is to collect intraocular pressure data with the EYEMATE pressure sensor in patients with BKPRO type and determine the relationship between the following glaucoma characteristics: intraocular pressure, characteristics and evolution of the optic nerve, visual fields, and OCT of the optic nerve. The intraocular pressure will be measured by three means. First, there will be mapping of the diurnal fluctuation of IOP with daily IOP self-measurement profiles with the EYEMATE system (subjects). Secondly, there will be mapping of fluctuation of IOP measurements with the EYEMATE system (site staff). Thirdly, the IOP will be evaluated through the measurement of the Schiotz tonometer on the limbal conjunctiva.

The primary performance objective is to collect IOP data with the EYEMATE system and compare the level of agreement between IOP measurements made using schiotz tonometry and the EYEMATE system over the first 24 months following implantation. The secondary performance objective is to determine the relationship between the IOP data with the use of the EYEMATE system and the progression of glaucoma through the evaluation of the characteristics of the optic nerve, visual fields, and OCT of the peripapillary retinal nerve fiber layers in patients with BKPRO type 1. The secondary safety objective is to evaluate the safety and tolerability of the EYEMATE pressure sensor, record adverse effects and incidence of device deficiencies in the first 24 months through the recording of incidence, nature, seriousness, severity and duration of adverse events at day 1 and at months 1, 4, 8, 12, 16, 20, 24 following implantation of the EYEMATE pressure sensor.

ELIGIBILITY:
Inclusion Criteria:

1. Keratoprosthesis surgery indicated, defined as having a severely opaque and vascularised cornea AND either a verifiable history of two or more prior failed corneal transplant procedures, limbal stem cells deficiency or a medical condition such as alkali burns or autoimmune disease that makes the success of a traditional corneal transplant procedure unlikely.
2. Ability and willingness to attend all scheduled visits and comply with all study procedures.

Exclusion Criteria:

1. Reasonable chance of success with traditional keratoplasty.
2. Current retinal detachment
3. Connective tissue diseases
4. History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to PRO-IOP implantation
5. History of ocular or periocular malignancy
6. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, or silicone (component of the device)
7. Presence of another active medical eye implant and/or other active medical implants in the head/neck region
8. Signs of current infection, including fever and current treatment with antibiotics
9. Severe generalized disease that results in a life expectancy shorter than a year
10. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
11. Currently pregnant or breastfeeding
12. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device
13. Intraoperative complication that would preclude implantation of the study device
14. Subject and/or an immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the contract research organization.
15. Previous or concurrent enrollment of the contralateral eye in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
IOP data gathering | 24 months
  • To collect IOP data with the PRO-IOP system and evaluate the performance of the PRO-IOP system in the first 24 months following implantation. This will be compared to digital palpation and tonopen.

SECONDARY OUTCOMES:
Relationship between IOP data and determinants factors of glaucoma | 24 months
  To determine the relationship between the IOP data with the use of the EyeMate system and the evolution of the other determinant factors of glaucoma through a correlation analysis of IOP with the characteristics and evolution of the optic nerve, visual fields, and OCT of the peripapillary retinal nerve fiber layers in patients with BKPRO type 1.
Safety and tolerability of the EyeMate sensor | 24 months
  To evaluate the safety and tolerability of the EyeMate pressure sensor and record adverse effects in the first 24 months through the recording of incidence, nature, seriousness, severity and duration of adverse events at day 1 and at months 1, 4, 8, 12, 16, 20, 24 following implantation of the PRO-IOP pressure sensor. Recording of incidence of device deficiencies at day 1 and at months 1, 4, 8, 12, 16, 20, 24 following implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Harissi-Dagher, MD, Principal Investigator — CHUM

IPD SHARING:
Plan to Share IPD: No